CLINICAL TRIAL: NCT00351559
Title: Invasive Monitoring Attenuation Through Gene Expression (IMAGE) Trial
Brief Title: IMAGE: A Comparison of AlloMap Molecular Testing and Traditional Biopsy-based Surveillance for Heart Transplant Rejection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XDx (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CA-0004
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Graft Rejection; Heart Diseases
Keywords: allograft; rejection; biopsy; gene; expression; cardiac; heart; transplant
MeSH Terms: conditions — Heart Diseases; Rejection, Psychology

INTERVENTIONS:
Device: AlloMap molecular expression testing
Procedure: Right ventricular endomyocardial biopsy

SUMMARY:
This study is designed to evaluate the safety and efficacy of a leukocyte gene expression profiling method in the monitoring of asymptomatic heart transplant patients for acute rejection.

DETAILED DESCRIPTION:
Cardiac allograft rejection is experienced by 20-50% of patients at least once during the first year after cardiac transplantation under the present immunosuppression regimens. With a higher incidence of acute cellular rejection (ACR) in the first six months post-transplant, ACR continues to occur beyond the first year post-transplant. However, the optimal strategy for detecting rejection during this period of lower risk period for ACR is still controversial. The standard for rejection surveillance has been the endomyocardial biopsy (EMB). However, EMB is invasive, causes morbidity, and is subject to sampling error and inter-observer variability.

Gene expression profiling (GEP), with its high negative predictive value (NPV) for acute cellular rejection (ACR), appears to be well suited to identify low-risk patients who can be safely managed without routine invasive endomyocardial biopsy (EMB).

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant recipients who are > 6 months to 5 years (> 6-60 months) post-transplant.
2. Age ≥ 18 years.
3. Stable outpatient being seen for routine monitoring of rejection. Stability is defined as absence of prior or current evidence of either severe cardiac allograft vasculopathy (CAV) or antibody-mediated rejection (AMR) with associated hemodynamic compromise.

   1. Severe CAV is defined as either

      * > 50% left main stenosis;
      * ≥ 50% stenosis in ≥ 2 primary vessels (proximal 1/3 or middle 1/3 of the LAD or LCx, RCA to takeoff of PDA in right-dominant coronary circulations) or
      * Isolated branch stenoses of > 50% in all 3 systems (diagonal branches, obtuse marginal branches, distal 1/3 of LAD or LCx, PDA, PLB, and RCA to takeoff of PDA in non-dominant systems).
   2. AMR with associated hemodynamic compromise is defined as AMR (defined according to local criteria) with either

      * A left ventricular ejection fraction (LVEF) ≤ 30% or at least 25% lower than the baseline value,
      * A cardiac index < 2 l/min/m2, or
      * The use of inotropic agents to support circulation.
4. Left ventricular ejection fraction ≥ 45% by Echocardiography, Multiple Gated Acquisition (MUGA) scan, or ventriculography at study entry (baseline / enrollment study).

Exclusion Criteria:

1. Patients < 7 calendar months after heart transplantation.
2. Any clinical signs of declining graft function:

   1. Symptoms of Congestive Heart Failure (CHF) at the enrollment visit.
   2. Signs of decompensated heart failure, including the development of a new S3 gallop at the enrollment visit.
   3. Elevated right heart pressures with diminished cardiac index < 2.2 L/min/m2 that is new compared to a previous measurement within 6 months.
   4. Decrease in LVEF as measured by echocardiography: ≥ 25% compared to prior measurement within 6 months.
3. Rejection therapy for biopsy-proven ISHLT Grade 3A or higher during the preceding 2 months.
4. Major changes in immunosuppression therapy within previous 30 days (e.g., discontinuation of calcineurin inhibitors, switch from mycophenolate mofetil to sirolimus or vice versa).
5. Unable to give written informed consent.
6. Patient receiving hematopoietic growth factors (e.g., Neupogen, Epogen) currently or during the previous 30 days.
7. Patients receiving ≥ 20 mg/day of prednisone equivalent corticosteroids at the time of enrollment.
8. Patient enrolled in a trial requiring routine surveillance endomyocardial biopsies.
9. Patient received transfusion within preceding 4 weeks.
10. Patients with end-stage renal disease requiring some form of renal replacement therapy (hemodialysis or peritoneal dialysis).
11. Pregnancy at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2005-01; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Time from study enrollment to the earliest date of decrease in left ventricle function (left ventricular ejection fraction [LVEF] decrease ≥ 25% from baseline)
Time from study enrollment to the development of clinically overt rejection (heart failure, hemodynamic compromise)
Time from study enrollment to death from any cause

SECONDARY OUTCOMES:
Number of deaths and cause of death
Number of biopsies planned and performed
Time to and number of biopsy-related complications, including bleeding, perforation and tamponade requiring pericardiocentesis, worsening of tricuspid regurgitation (TR) by 1 grade above 2+ or new TR at least 3+ or greater

CONTACTS AND LOCATIONS:
Overall Officials: Hannah A Valantine, MD, MRCP, FACC, Study Chair — Stanford University; Michael Pham, MD, MPH, Principal Investigator — VA Palo Alto Health Care System; Mario C Deng, MD, Principal Investigator — Columbia University, New York Presbyterian Hospital; Jeffrey J Teuteberg, MD, Principal Investigator — University of Pittsburgh Medical Center; A G Kfoury, MD, Principal Investigator — Intermountain Medical Center; Dale G Renlund, MD, Principal Investigator — Intermountain Medical Center; Randall C Starling, MD, MPH, Principal Investigator — The Cleveland Clinic; Allen Anderson, MD, Principal Investigator — University of Chicago; Thomas Cappola, MD, ScM, Principal Investigator — University of Pennsylvania; Andrew Kao, MD, Principal Investigator — Mid America Heart Institute - St. Luke's Hospital; William G Cotts, MD, Principal Investigator — Northwestern University; Roberta C Bogaev, M.D., FACC, FACP, Principal Investigator — Texas Heart Institute at St. Luke's Episcopal Hospital; David Baran, MD, Principal Investigator — Newark Beth Israel Medical Center; Greg Ewald, MD, Principal Investigator — Barnes-Jewish Hospital
Locations (13):
- United States (13):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Mid America Heart Institute - St. Luke's Hospital, Kansas City, Missouri
  - Barnes Jewish Hospital - Washington University, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University Medical Center - New York Presbyterian Hospital, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah

REFERENCES:
- [Background] Deng MC, Eisen HJ, Mehra MR, Billingham M, Marboe CC, Berry G, Kobashigawa J, Johnson FL, Starling RC, Murali S, Pauly DF, Baron H, Wohlgemuth JG, Woodward RN, Klingler TM, Walther D, Lal PG, Rosenberg S, Hunt S; CARGO Investigators. Noninvasive discrimination of rejection in cardiac allograft recipients using gene expression profiling. Am J Transplant. 2006 Jan;6(1):150-60. doi: 10.1111/j.1600-6143.2005.01175.x. PMID 16433769
- [Background] Evans RW, Williams GE, Baron HM, Deng MC, Eisen HJ, Hunt SA, Khan MM, Kobashigawa JA, Marton EN, Mehra MR, Mital SR. The economic implications of noninvasive molecular testing for cardiac allograft rejection. Am J Transplant. 2005 Jun;5(6):1553-8. doi: 10.1111/j.1600-6143.2005.00869.x. PMID 15888068
- [Background] Marboe CC, Billingham M, Eisen H, Deng MC, Baron H, Mehra M, Hunt S, Wohlgemuth J, Mahmood I, Prentice J, Berry G. Nodular endocardial infiltrates (Quilty lesions) cause significant variability in diagnosis of ISHLT Grade 2 and 3A rejection in cardiac allograft recipients. J Heart Lung Transplant. 2005 Jul;24(7 Suppl):S219-26. doi: 10.1016/j.healun.2005.04.001. PMID 15993777
- [Background] Pham MX, Deng MC, Kfoury AG, Teuteberg JJ, Starling RC, Valantine H. Molecular testing for long-term rejection surveillance in heart transplant recipients: design of the Invasive Monitoring Attenuation Through Gene Expression (IMAGE) trial. J Heart Lung Transplant. 2007 Aug;26(8):808-14. doi: 10.1016/j.healun.2007.05.017. PMID 17692784
- [Derived] Deng MC, Elashoff B, Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Shahzad K, Hiller D, Yee J, Valantine HA; IMAGE Study Group. Utility of gene expression profiling score variability to predict clinical events in heart transplant recipients. Transplantation. 2014 Mar 27;97(6):708-14. doi: 10.1097/01.TP.0000443897.29951.cf. PMID 24637869
- [Derived] Pham MX, Teuteberg JJ, Kfoury AG, Starling RC, Deng MC, Cappola TP, Kao A, Anderson AS, Cotts WG, Ewald GA, Baran DA, Bogaev RC, Elashoff B, Baron H, Yee J, Valantine HA; IMAGE Study Group. Gene-expression profiling for rejection surveillance after cardiac transplantation. N Engl J Med. 2010 May 20;362(20):1890-900. doi: 10.1056/NEJMoa0912965. Epub 2010 Apr 22. PMID 20413602
- See also: Sponsor's web site — http://www.xdx.com